CLINICAL TRIAL: NCT03572491
Title: A Phase 3, an Open Clinical Trials to Evaluate Effectiveness, Safety and Immunogenicity of a Allantoic Split Inactivated Seasonal Influenza Vaccine in Healthy Adults
Brief Title: Preventive Effectiveness, Safety and Immunogenicity of a Allantoic Split Inactivated Seasonal Influenza Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Research Institute for Biological Safety Problems (Other Government)
Collaborators: Asfendiyarov Kazakh National Medical University (Other); Research Institute of Influenza, Russia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VSI-III-01/2017
Record Dates: First submitted 2018-06-05; First posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Human Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: The main group - group 1 = 1000 volunteers will be vaccinated with the vaccine "Allan-toxin split inactivated against seasonal influenza vaccine".
  In the main group, a subgroup will be singled out - a group of 1a = 200 volunteers who will be examined for safety, immunogenicity and immunity.
  The observation group is a group of 2 = 1000 people who, when confirming the diagnosis of influenza, will compare the incidence with the main group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allantoic split inactivated seasonal influenza vaccine (Experimental): A allantoic split inactivated seasonal influenza vaccine has been prepared on eggs and is made from inactivated parts of the following influenza virus strains: NYMC X-275 (A/PR/8/34 (M, PB2, PA, NS, NP genes) и A/Michigan/45/2015 (PB1, HA, NA genes)), NYMC X-263В (A/PR/8/34 (PB1, PB2, PA, NS, NP, М genes) и A/Hong Kong/4801/2014 (HA, NA genes)), NYMC BX-35 (B/Lee/40 (NP gene), B/Panama/45/90 (PB2, М genes) и B/Brisbane/60/2008 (HA, NA PB1, PA, NS genes)).
  Interventions: Biological: influenza vaccine

INTERVENTIONS:
Biological: influenza vaccine — Allantoic split inactivated seasonal influenza vaccine

SUMMARY:
The study is Multicenter, phase 3, Open-Label trial that explored the preventive effectiveness, safety and immunogenicity of single dose a allantoic split inactivated seasonal influenza vaccine in healthy adults.

DETAILED DESCRIPTION:
The study will include 2000 volunteers, 1,000 of whom will be vaccinated intramuscularly with a single dose of allantoic split inactivated seasonal influenza vaccine.

All participants will be observed for 6 months to evaluate the effectiveness of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both sexes aged from 18 years.
* Literate and willing to provide written informed consent.
* A signed informed consent.
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Allergic reactions to chicken proteins, or any preceding vaccination.
* Acute illness with a fever (37.0 C).
* Vaccination against influenza in the 2017/2018 season.
* Current or recent (within two weeks of enrollment) acute respiratory illness with or without fever.
* Hypersensitivity after previous administration of any vaccine.
* History of chronic alcohol abuse and/or illegal drug use.
* A positive pregnancy test for all women of childbearing potential.
* Administration of immunosuppressive drugs or other immune modifying drugs within 4 weeks prior to study enrollment.
* Acute or chronic clinically significant pulmonary disease, cardiovascular disease, gastrointestinal disease, liver disease, neurological illness, liver disease, blood disease, skin disorder, endocrine disorder, neurological illness and psychiatric disorder as determined by medical history, physical examination or clinical laboratory screening tests, which in the opinion of the investigator, might interfere with the study objectives.
* History of leukemia or any other blood or solid organ cancer.
* Receipt of antivirals, antibiotics, immunoglobulins or other blood products within 4 weeks prior to study enrollment or planned receipt of such products during the period of subject participation in the study.
* Participation in another clinical trial within the previous three months or planned enrollment in such a trial during the period of this study.
* Subjects who are, in the opinion of the investigator, at significantly increased risk of non-cooperation with requirements of the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Preventive efficacy - Incidence of influenza among vaccinated and unvaccinated volunteers | 180 days
  An assessment of the incidence of influenza among vaccinated and unvaccinated volunteers will be conducted within 180 days of observation (PCR diagnostics for the detection of influenza viruses).

SECONDARY OUTCOMES:
Percentage of Participants With Solicited Local and Systemic Adverse Events (AEs) | 21 days
  Participants recorded solicited injection site and systemic adverse events in a Subject Diary. Solicited Locals AEs were: Injection Site Pain, Injection Site Redness, Injection Site Swelling, Injection Site Induration and Injection Site Ecchymosis. Solicited Systemic AEs were: Pyrexia, Malaise, Chills, Fatigue, Headache, Sweaty, Myalgia, Arthralgia, Nausea and Vomiting.
Percentage of Participants Reporting One or More Treatment-emergent Adverse Events (TEAE) | Greater than 2 hours after administration of any dose of vaccine or placebo through 7 days following any dose
Percentage of Participants With Abnormal Safety Laboratory Tests at Least Once Post Dose Reported as AEs | Greater than 2 hours after administration of any dose of vaccine or placebo through 7 days
Serious adverse events (SAEs), including abnormal laboratory findings | up to 24 weeks
Geometric Mean Fold Increase in HI Antibody Titer | Change from Baseline HI Antibody Titer at 21, 90 and 180 days
  1A group
Seroconversion Rate of Hemagglutination Inhibition (HI) Antibody Titer | Change from Baseline HI Antibody Titer at 21, 90 and 180 days
  1A group - Seroconversion rate was measured by hemagglutination inhibition (HI) antibody titer for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21, 90, 180 days after vaccination. Seroconversion rate was defined as the percentage of participants achieving a minimal 4-fold increase from the Baseline HI antibody titer in participants with a Baseline titer ≥10, or achieving an HI antibody titer of ≥40 in participants with a Baseline titer <10.
Seroprotection Rate of HI Antibody Titer | Change from Baseline HI Antibody Titer at 21, 90 and 180 days
  Seroprotection rate, defined as the percentage of participants with HI antibody titer of ≥40, was measured by HI antibody titer for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21, 90, 180 days after vaccination. Day 1 data is reported for reference.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute for Biological Safety Problems, Gvardeysky, Jambul, Kazakhstan

IPD SHARING:
Plan to Share IPD: No